CLINICAL TRIAL: NCT04904757
Title: Willingness of Women to Undergo a Contrast-enhanced Spectral Mammography (CESM) for Breast Cancer Screening and Their Experience Before and After CESM
Brief Title: Contrast-enhanced Spectral Mammography (CESM) Breast Cancer Screening
Acronym: S-CESM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Matthew Miller, MD PhD, Radiology-Breast Imaging Faculty, Clinical Assistant Professor, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB#18853
Record Dates: First submitted 2021-02-26; First posted 2021-05-27 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Mammographic Breast Density; Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CESM Pre and Post Survey (Other): Subject will be asked to complete a questionnaire that will ask you about your general attitude toward Contrast-Enhanced Spectral Mammography (CESM). Questions will include:
  * Thoughts regarding risk of breast cancer
  * Concerns regarding contrast procedures such as the CESM
  * Past mammogram/breast imaging experience
  Interventions: Device: Contrast-enhanced spectral mammography (CESM)

INTERVENTIONS:
Device: Contrast-enhanced spectral mammography (CESM) — CESM is a mammogram performed after the injection of IV contrast. CESM is used most often when additional information is needed after a standard mammogram. CESM has also been used to determine the extent of a known breast cancer, to screen patients at high risk for developing breast cancer due to a family history or positive cancer genes, and for women with dense breast tissue. Two images are taken almost at the same time during the exam, after the iodine based contrast injection is administered. The first image is comparable to a regular mammogram. The second image shows areas that take up the contrast (enhance) showing increased blood flow. Breast cancers often enhance with contrast due to a greater amount of blood vessels. Non-cancerous lesions can also have greater blood flow.

SUMMARY:
The purpose of this study is to evaluate how well women may adopt a Contrast-enhanced Spectral Mammography (CESM) as their yearly breast screening test compared to the standard 2-D or 3-D mammogram.

DETAILED DESCRIPTION:
Contrast-enhanced spectral mammography (CESM) is an FDA approved tool for breast cancer detection. However, adoption into clinical practice has been slow. In this study, we will explore patient issues related to the use of CESM for breast cancer screening. For this study, 210 women with heterogeneous or dense breast tissue reported on a previous mammogram, will be recruited to undergo a screening Contrast-enhanced Spectral Mammography (CESM). The CESM will serve as the subject's annual screening breast exam for clinical care. A survey will be administered before and after the examination that evaluates the patient experience. Women will not be at high risk for breast cancer (<20% lifetime risk). All abnormal findings will be acted upon independently. Results of the general screening population survey will be compared with those of women who choose to undergo the CESM examination in order to evaluate the influence of age, education, and lifetime risk on decision making about advanced screening.

ELIGIBILITY:
Inclusion Criteria:

* • Female

  * 40 to 69 years
  * Previous normal mammogram (BI-RADS 1 or 2) showing heterogeneous or extremely dense breast tissue within last 24 months
  * Scheduled for screening mammogram as part of the patient's clinical care

Exclusion Criteria:

* • No mammogram within last 24 months

  * Fatty or scattered fibroglandular tissue on last mammogram
  * History of allergy to iodinated contrast
  * History of renal disease or renal function abnormalities
  * Pregnant women
  * History of diabetes
  * History of paraproteinemia syndromes such as multiple myeloma
  * History of collagen vascular disease
  * History of vascular disease (coronary artery disease, myocardial infarction, carotid disease, peripheral vascular disease, or known visceral artery disease)
  * Previously identified as high risk for breast cancer (>20% lifetime risk)
  * Asthma
  * Sickle Cell Anemia
  * Currently on Dialysis

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 210 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the patient experience during a screening CESM | 16 months
  Plan for primary variable analysis: To evaluate the patient experience during a screening CESM to better understand if women find the experience of contrast injection to be too invasive or unpleasant to repeat or recommend to a friend.
  Data summarization: Pre and post CESM survey responses that are binary or Likert scaled responses will be summarized by frequencies and percentages. Pre and post CESM survey responses that are continuous scaled responses will be summarized by the mean and standard deviation, the median and interquartile range, and the range of distribution.

SECONDARY OUTCOMES:
determine if there is an association between the willingness to undergo CESM and age, level of education, and breast cancer related risk factors. | 16months
  We will evaluate differences by age, education, and risk factors as to whether these drive willingness to undergo CESM.
  Data summarization: Binary risk factors will be summarized by frequencies and percentages. Continuous scaled risk factors will be summarized by the mean and standard deviation, the median and interquartile range, and the range of distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- UVA Breast Care Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04904757/Prot_000.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04904757/ICF_001.pdf